CLINICAL TRIAL: NCT04215003
Title: This is a Phase Ib/II, Prospective , Open-label, Single Center, Bayesian Adaptive Design, Umbrella Study Evaluating the Efficacy and Safety of Neo-adjuvant Therapy in Patients With Breast Cancer.
Brief Title: A Clinical Trial of Breast Cancer Neo-adjuvant Therapy Based on Molecular Pathway in FUSCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Precision neo-adjuvant therapy of Breast Cancer Based on Molecular pathway, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC0N026
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; neo-adjuvant therapy; molecular pathway; umbrella trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Active Comparator): 6 cycles of Paclitaxel,Carboplatin, Herceptin and Pertuzumab treatment with a good clinical benefit response depending on HR/HER-2 status.
  Interventions: Drug: A
- B (Experimental): 2 cycles of Paclitaxel,Carboplatin, Herceptin treatment with a good clinical benefit response depending on HR/HER-2 status following surgery
  Interventions: Drug: B
- CL4 (Experimental): HR+ and HER2-; No correlated pathway variation
  Interventions: Drug: CL4

INTERVENTIONS:
Drug: A — Paclitaxel: paclitaxel 80 mg/m2 ivgtt d1, d8, d15, 28 days per cycle. Carboplatin: carboplatin AUC=2 ivgtt d1, d8, d15, 28 days per cycle. Herceptin: 4 mg/kg (loading dose 8mg/kg) ivgtt d1,8,15, 22, 28 days per cycle,6 cycles.
  Pertuzumab: 420-mg ( loading dose 840mg) ivgtt d1, 21 days per cycle,6 cycles.
  Arms: A
Drug: B — Paclitaxel: paclitaxel 80 mg/m2 ivgtt d1, d8, d15, 28 days per cycle. Carboplatin: carboplatin AUC=2 ivgtt d1, d8, d15, 28 days per cycle.
  Arms: B
Drug: CL4 — SHR6390（CDK4/6 inhibitor）125 mg qd(three week on one week off); oral letrozole 2.5 mg daily； Adebrelimab was given intravenously, 600mg each time, once every 2 weeks; Premenopause：Goserelin 3.6mg IM IM Q4W.
  Arms: CL4

SUMMARY:
This is a Phase Ib/II, prospective , open-label, single center, Bayesian adaptive design, umbrella study evaluating the efficacy and safety of neo-adjuvant therapy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old Expected survival > 12 months Baseline ECOG Performance Status rating 0-1 Naïve to chemotherapy or hormonal treatments Radiologically confirmed and biopsy diagnosed invasive ductal carcinoma of breast and prepared to be treated surgically Locally advance breast cancer of stage IIb-IIIc No concurrent malignancy (except controlled cervical carcinoma in situ or basal cell carcinoma of skin) Patients have measurable lesions (according to RECIST v1.1 criteria) Intention to cooperate with baseline puncture and neoadjuvant therapy No advanced metastasis or metastasis involving brain or liver Adequate bone marrow function, blood routine examination shows neutrophil count ≥ 1.5x109/L, hemoglobin level ≥ 100 g/L, Platelets ≥ 100 x 109/L Adequate liver and kidney function, serum aminotransferase (AST) ≤ 60U/L, serum total bilirubin ≤ 2.5 times ULN, serum creatinine ≤110μmol/L, urea nitrogen ≤7.1mmol/L No coagulation abnormality Normal heart function, with normal ECG and LVEF ≥ 55% Women of childbearing age agree to take reliable contraceptive measures during clinical trials, and negative serum or urine pregnancy test within 7 days prior to administration No coagulation abnormality Sign the informed consent statement and voluntarily receive follow-ups, treatments, laboratory tests and other research procedures according to protocol.

Exclusion Criteria:

* Previous regional or systemic treatment for breast cancer (include but not limited to chemotherapy, radiotherapy, targeted therapy, other clinical trials) Inflammatory breast cancer, bilateral breast cancer or breast cancer already with distant metastasis Complicated with uncontrolled lung disease, severe infection, active peptic ulcer, blood clotting disorders, severe uncontrolled diabetes, connective tissue disorders or bone marrow suppression, and intolerance to neoadjuvant therapy or related treatment Peripheral neuropathy >1 degree caused by any reason History of congestive heart failure, uncontrolled or symptomatic angina, arrhythmias or history of myocardial infarction, refractory hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg); Breast cancer during lactation or pregnancy Unwillingly to receive baseline puncture or neoadjuvant therapy Mental illness or incompliance to treatment caused by other reasons Known history of severe hypersusceptibility to any agents used in the treatment protocol Patients received major surgery or suffered from severe trauma within 2 months of first administration Currently enroll or recently used (30 days within enrollment) other agent under research or involved in other trial Known to be infected with human immunodeficiency virus (HIV) Other circumstances considered to be inappropriate to be enrolled by researchers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pathologic Complete Response (pCR) | through study completion, up to 24 weeks
  pCR is defined as the absence of noninvasive tumor residuals in breast and axillary lymph nodes (ypT0/is ypN0) after neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 weeks
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shao Zhimin, Shanghai, Please Select
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided